CLINICAL TRIAL: NCT06662864
Title: Study on Sleep, Lifestyle and Quality of Life in Women With Breast Cancer Undergoing Endocrine Therapy
Brief Title: Study on Sleep, Lifestyle and Quality of Life in Women With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Institut Rafael (Other)
Responsible Party: Sponsor
Other Study IDs: IR-2024-002; 2024-A01086-41 (Other: ID-RCB)
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancers
Keywords: breast cancer; endocrine therapy; Quality of Life; anxiety and depression; integrative medecine; sleep disorders
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Depression; Sleep Wake Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: women aged 20 to 85 years old diagnosed with hormone receptor positive breast cancer
  Interventions: Other: Patients reported outcomes; Other: questionnaire global Pittsburgh Sleep Quality Index (PSQI)

INTERVENTIONS:
Other: Patients reported outcomes — Patients reported outcomes were collected via telephone
  Other Names: survey; questionnaires
Other: questionnaire global Pittsburgh Sleep Quality Index (PSQI) — Patients reported outcomes were collected via telephone

SUMMARY:
This was a prospective survey conducted at a single site, the Rafaël Institute, France. Eligible patients were women aged 20 to 85 years old diagnosed with hormone receptor positive breast cancer and undergoing adjuvant endocrine therapy since at least 3 months. Patients reported outcomes were collected via telephone. Primary endpoint consisted in the global Pittsburgh Sleep Quality Index (PSQI). Secondary endpoints included evaluation of anxiety and depression (hospital anxiety and depression scale, HADS), pain (numeric rating scale), health related quality of life (EQ-5D-5L) and lifestyle habits (questionnaire designed for this study). Descriptive statistical analyses were performed with the intention to treat population.

Sixty patients were included after providing oral informed consent. The PSQI evaluation of subjective sleep quality revealed a global score of 7.40. The majority of patients (73.3%) obtained a score > 5. Among those, 50% obtained a score between 6 and 10, while 23.3% had a score between 11 and 15. In contrast, only 26.7% of patients were good sleepers with a score <=5. Mean scores for anxiety and depression were 6.5 (+/- 3.8) and 3.3 (+/- 3.2) indicating non cases. The majority of patients (44; 73%) said to suffer from joint pain. In a matrix correlation test, the correlation index of PSQI with anxiety, depression and pain were +0.19, +0.28 and +0.44, respectively. The mean score in the EQ-5D-5L visual analogue scale was 63.0 (+/-13) for the entire sample. 44% of patients reported to use complementary medicine to help them feel better.

The majority of patients with breast cancer undergoing endocrine therapy were considered poor sleepers. Pain was moderately correlated with sleep disorders while both anxiety and depression showed a weak correlation. Awareness and knowledge on integrative approaches to support and improve patients' outcomes remains low among breast cancer patients.

DETAILED DESCRIPTION:
Adjuvant therapy with either tamoxifen or aromatase inhibitors reduces breast cancer recurrence and improves overall survival in patients with hormone receptor-positive breast cancer. However, the benefits achieved with adjuvant endocrine therapy come at a cost. A variety of negative symptoms can substantially impair patients' quality of life and treatment adherence. Sleep disorder, a well-known side effect of endocrine therapy, may compromise treatment effectiveness and serves as relevant behavioral marker of poor prognosis. In order to be able to offer personalized solutions combining conventional pharmacological medicine with non-pharmacological approaches, it is important to understand the impact of the sleep disorders particularly in women with breast cancer on endocrine therapy who present an increased risk of insomnia. The primary aim of this study was to assess sleep quality and its relationship with anxiety, depression and pain. Patients' lifestyle, knowledge on integrative approaches to health and global quality of life were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were women aged 20 to 85 years old diagnosed with hormone receptor positive breast cancer and undergoing adjuvant endocrine therapy since at least 3 months

Exclusion Criteria:

* less than 18 years old

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 20 to 85 years old diagnosed with hormone receptor positive breast cancer and undergoing adjuvant endocrine therapy since at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
questionnaire Pittsburgh Sleep Quality Index (PSQI) | 30 minutes
  The PSQI comprises 19 self-rated questions grouped into 7 components (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction). Each component score weighs equally on a 0 (no difficulty) to 3 (severe difficulty). The scores of 7 components are summed up to a global PSQI score, which ranged from 0 to 21 points with a cutoff score of ≤ 5 indicating good sleep quality.

SECONDARY OUTCOMES:
hospital anxiety and depression scale, HADS | 30 minutes
  HADS consisted of 14 items. Seven of the items indicate anxiety and the remaining seven items indicate depression. The answer format offers four response options, which are scored with values ranging from 0 to 3. This results in scale values between 0 and 21 for each scale. The original test authors defined three ranges for both of the scales: 0-7 (non-cases), 8-10 (doubtful cases), and 11-21(cases).
pain scale (numeric rating scale) | 30 minutes
  numeric rating scale of 0 to 10 where zero means "no pain" and ten means "the worst possible pain"
questionnaire health related quality of life EQ-5D-5L | 30 minutes
  The EQ-5D-5L score is presented between 0 (worst imaginable health) and 100 (best imaginable health) for their current overall health-related quality of life.
questionnaire lifestyle habits | 30 minutes
  Questions designed for this study

CONTACTS AND LOCATIONS:
Locations (1):
- Institute Rafaël, Levallois-Perret, Institut Rafael, France

IPD SHARING:
Plan to Share IPD: No